CLINICAL TRIAL: NCT04655742
Title: A Prospective, Multi-center, Single-arm Clinical Investigation for Evaluation of the Safety and Effectiveness of the MicroPort™ CardioFlow VitaFlow™ Transcatheter Aortic Valve System in the Treatment of Severe Aortic Stenosis
Brief Title: VitaFlow™ Transcatheter Aortic Valve System Pre-market Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai MicroPort CardioFlow Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: valve-2014-04
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm, treatment group (Experimental): Subjects in the treatment group will be implanted with the VitaFlow™ Transcatheter Aortic Valve System
  Interventions: Device: VitaFlow™ Transcatheter Aortic Valve System

INTERVENTIONS:
Device: VitaFlow™ Transcatheter Aortic Valve System — VitaFlow™ Transcatheter Aortic Valve System contains a valve stent-VitaFlow™ Aortic Valve, a delivery system-VitaFlow™ Delivery System,loading tools, a balloon dilatation catheter, and an introducer set

SUMMARY:
This is a pre-market clinical investigation aiming to evaluate the safety and effectiveness of MicroPort™ CardioFlow VitaFlow™ Transcatheter Aortic Valve System for the treatment of severe aortic stenosis.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm clinical investigation for evaluation of the safety and effectiveness of the MicroPort™ CardioFlow VitaFlow™ Transcatheter Aortic Valve System in the Treatment of Severe Aortic Stenosis. The investigation has two phases.

Phase I（FIM）：The FIM stage is a prospective, multicenter, single-arm observational clinical investigation, aiming to evaluate the feasibility and safety of the MicroPort™ CardioFlow VitaFlow™ Transcatheter Aortic Valve System. A total of 10 patients will be enrolled and 30-day clinical outcomes will be collected.

Phase II (Pivotal)：The pivotal stage is a prospective, multi-center, single-arm clinical investigation with the performance goal, aiming to evaluate the safety and effectiveness of MicroPort™ CardioFlow VitaFlow™ Transcatheter Aortic Valve System for the treatment of severe aortic stenosis. A total of 110 patients will be enrolled in 11 clinical centers across China. Clinical or telephone follow-up is scheduled at 30 days, 6 months, 12 months, and 2 to 5 years annually post-procedure.

ELIGIBILITY:
Inclusion criteria :

Enrollment was limited to patients who met all of the following criteria:

1. Age ≥ 70 years old(Phase II)/Age ≥18 years old,male or female who are not pregnant (Phase I);
2. Patients have severe aortic stenosis: Mean gradient> 40mmHg(1mmHg = 0.133kPa), or peak velocity> 4m/s, or an aortic valve area(AVA) <1.0 cm² (or AVA index <0.6 cm²/m²);
3. NYHA classification ≥ II;
4. Life expectancy> 12 months;
5. Anatomically suitable for transcatheter aortic valve implantation;
6. Assessed by a multidisciplinary heart team as a patient unsuitable for surgical aortic valve replacement;
7. Patients who can understand the purpose of the investigation, volunteer to participate in and sign the informed consent form, and are willing to comply with relevant examinations and follow-up visits.

Exclusion criteria:

1. Acute myocardial infarction occurred within 30 days before the treatment;
2. Patients with congenital unicuspid aortic valve or aortic root anatomy and lesions that are not suitable for transcatheter valve implantation;
3. Any therapeutic heart surgery within 30 days;
4. Mixed aortic valve disease(aortic stenosis with severe regurgitation); moderate and severe mitral stenosis; severe mitral regurgitation; severe tricuspid regurgitation;
5. Blood dyscrasia, including neutropenia (WBC < 3 × 10^9/L), acute anemia(HB <90 g/L), thrombocytopenia(PLT <50 × 10^9/L), hemorrhagic constitution, and coagulopathy disease;
6. Untreated coronary artery disease requiring revascularization;
7. Hemodynamic instability requiring systolic support or mechanical heart assistance;
8. Need for emergency surgery for any reason;
9. Obstructive hypertrophic cardiomyopathy;
10. Severe left ventricular dysfunction, left ventricular ejection fraction(LVEF) < 20%; severe pulmonary hypertension and right ventricular dysfunction;
11. Echocardiography suggests the presence of intracardiac masses, thrombi, or neoplasms;
12. Active peptic ulcer or history of upper gastrointestinal bleeding within 3 months;
13. Allergy to aspirin, heparin, ticlopidine, clopidogrel, nitinol, or contrast agents;
14. Cerebrovascular events including transient ischemic attack(TIA) occurred within 6 months;
15. Renal insufficiency decompensation(end creatinine clearance < 20ml/min), and / or end-stage renal disease require long-term dialysis treatment;
16. Vascular diseases affecting device access;
17. Active infectious endocarditis or other active infection;
18. Participated in clinical investigations of other drugs or medical devices before the election, and had not completed the primary endpoint;
19. The investigator judged that the patient had poor compliance and could not complete the study as required.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of device success-Phase I | at immediate post-procedure
All-cause mortality at 12 months post implantation-Phase II | at 12 months post-procedure

SECONDARY OUTCOMES:
Rate of major adverse events -Phase I | at 30 days post implantation
Hemodynamic performance-Phase II | at immediate post-procedure, discharge, 30 days, 6 months, 1 year and annually up to 5 years post implantation
  Hemodynamic performance, including the mean prosthetic valve gradient(in mmHg), the Effective orifice(in cm^2), and the degree of prosthetic valve regurgitation measured by transthoracic echocardiography (TTE)
Heart function(NYHA)-Phase II | at immediate post-procedure, discharge, 30 days, 6 months, 1 year and annually up to 5 years post implantation
Rate of safety events according to VARC2-Phase II | at immediate, 30 days, 1 year and annually up to 5 years post implantation
Rate of major cardiovascular and cerebrovascular events(MACCE)-Phase II | at immediate, 30 days, 1 year and annually up to 5 years post implantation
Rate of balloon pre-dilatation success-Phase II | at immediate post implantation
Rate of balloon post-dilatation success-Phase II | at immediate post implantation

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang